CLINICAL TRIAL: NCT05258539
Title: Breast Cancer Prevention and Screening Membership
Acronym: AdDePi_KS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP211502; 2021-A02665-36 (Other: ANSM)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Compliance; Risk Assessment; Cancer Risk Management Platform
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women aged 18 to 85 years who come to the CRMP for a breast cancer risk assessment. (Experimental)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Telephone calls at 2, 3 and 5 years with :
  * Lifestyle follow-up questionnaire.
  * Satisfaction questionnaire.

SUMMARY:
The AdDePi-KS project aims to contribute to the renovation of the breast cancer screening program. In order to improve information to women on breast cancer risk factors and their participation in organized screening, but also to reduce the incidence of the disease, the prevention policy currently in place could be adapted and optimized based on the assessment of women's individual risk factors.

The current principle of the platform is to offer women a breast cancer risk assessment and prevention consultation with a clinical examination and the use of three breast cancer risk calculation models: Tyrer Cuzick (TC) Mammorisk© (MMR) and CANRISK. In parallel to the use of these three softwares, the Eisinger and Manchester scores are also calculated to evaluate the indication of an oncogenetic consultation. At the end of this analysis, a personalized prevention plan (PPP) proposal, adaptable by the practitioner by shared decision with the consultant, is generated and proposed. The risk assessment and the monitoring strategy are explained to the consultant and when "actionable" risk factors are identified, personalized assistance is proposed (dietary consultation, smoking consultation, distribution of information documents, particularly on physical activity).

The objective of this study is to evaluate the impact of the consultation in the long term, in particular on compliance with the recommended monitoring methods and on the "actionable" personal risk factors. For this purpose, investigators propose to set up follow-up questionnaires at 2, 3 and 5 years. These questionnaires will also make it possible to monitor over time how the notion of risk is perceived and how this could influence primary (action on risk factors) and secondary (screening) prevention behaviors. Thus, by accompanying the objectives and methods of prevention in a genuine health democracy process, investigators will be able to identify certain obstacles and levers linked to the implementation of these actions.

DETAILED DESCRIPTION:
The AdDePi-KS project aims to contribute to the renovation of the breast cancer screening program. In order to improve information to women on breast cancer risk factors and their participation in organized screening, but also to reduce the incidence of the disease, the prevention policy currently in place could be adapted and optimized based on the assessment of women's individual risk factors. This approach would promote the implementation of measures that allow women to take a more active part in the decision-making process.

The current principle of the Cancer Risk Management Platform (CRMP) is to offer women a breast cancer risk assessment and prevention consultation with a clinical examination and the use of three breast cancer risk calculation models: Tyrer Cuzick (TC), Mammorisk© (MMR) and CANRISK. In parallel to the use of these three softwares, the Eisinger and Manchester scores are also calculated to evaluate the indication of an oncogenetic consultation. At the end of this analysis, a personalized prevention plan (PPP) proposal, adaptable by the practitioner by shared decision with the consultant, is generated and proposed. The risk assessment and the monitoring strategy are explained to the consultant and when "actionable" risk factors are identified, personalized assistance is proposed (dietary consultation, smoking consultation, distribution of information documents, particularly on physical activity).

The objective of this study is to evaluate the impact of the consultation in the long term, in particular on compliance with the recommended monitoring methods and on the "actionable" personal risk factors. For this purpose, investigators propose to set up follow-up questionnaires at 2, 3 and 5 years. These questionnaires will also make it possible to monitor over time how the notion of risk is perceived and how this could influence primary (action on risk factors) and secondary (screening) prevention behaviors. Thus, by accompanying the objectives and methods of prevention in a genuine health democracy process, investigators will be able to identify certain obstacles and levers linked to the implementation of these actions. Investigators believe that this approach will improve their understanding of the appropriation and dissemination of prevention practices for a better approach.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18-85 years who comes to the Cancer Risk Management Platform (CRMP) for a breast cancer risk assessment
* A woman who has signed an informed consent form
* Woman who is a beneficiary or entitled person of a social security plan

Exclusion Criteria:

* Woman diagnosed with breast cancer
* Woman under legal protection (guardianship, curatorship)
* Woman under AME

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with a compliance to the Personalized Prevention Plan established during the initial risk assessment consultation. | Compliance will be measured at 2, 3 and 5 years from the initial risk assessment consultation
  Modification of at least one behavior of the women with respect to certain actionable risk factors: alcohol consumption, overweight, sedentary lifestyle, smoking, fiber consumption.

SECONDARY OUTCOMES:
Proportion of participants with weight loss when overweight was identified at the initial risk assessment visit | 2, 3 and 5 years from the initial risk assessment consultation
Proportion of participants who were active in sports when no sports were identified at the initial risk assessment visit | at 2, 3 and 5 years
Proportion of participants who quit smoking | at 2, 3 and 5 years
Proportion of participants who changed their alcohol consumption when it was excessive at the initial risk assessment visit | at 2, 3 and 5 years
Proportion of participants who changed their diets when an imbalance in diet was noted at the initial risk assessment visit | at 2, 3, and 5 years
Proportion of women who completed their screening as recommended following the CRMP consultation | at 2, 3 and 5 years
Proportion of women's satisfaction with the initial consultation | at 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine UZAN, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.